CLINICAL TRIAL: NCT03905278
Title: Children Facing Parental Cancer : a Randomized Controlled Study Evaluating the Efficacy of a Psychological Intervention to Support Parenting
Brief Title: Parental Support Intervention in the Oncological Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aurore Liénard (Other)
Collaborators: Centre de Psycho-Oncologie (CPO) (Other); Erasme University Hospital (Other); Jules Bordet Institute (Other); Université Libre de Bruxelles (Other)
Responsible Party: Sponsor-Investigator, Aurore Liénard, Aurore Lienard, Coordinator of the Psycho-Oncology Clinic at the Bordet Institute, Université Libre de Bruxelles
Organization: Université Libre de Bruxelles (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CE2681
Record Dates: First submitted 2019-01-22; First posted 2019-04-05 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Parent-Child Relations; Parenting; Communication Programs
Keywords: parental cancer; parental guidance; parent-child communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: The effectiveness of the parental support intervention is assessed through a longitudinal two arms, randomized controlled trial and the experimental condition, the two significant caregivers of the children or the individual caregiver receive the intervention composed of an informational booklet and a psychological intervention. In the control condition, the participants receive the informational booklet before being registered in a waiting list for the psychological intervention. The intervention should ideally last two months. Assessments are conducted at two periods : before and after the intervention for the experimental group and at 9 weeks of interval for the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental guidance (Experimental): In the experimental condition, the two significant caregivers of the child or the individual caregiver receive the intervention composed of an informational booklet and a psychological intervention. The intervention consists of four sessions, centered on supporting the child in the context of parental cancer principally through communication.
  Assessments are conducted at two periods : before and after the intervention.
  Interventions: Behavioral: Parental guidance
- Waiting List group (No Intervention): In the control condition, the participants receive the informational booklet before being registered in a waiting list for the psychological intervention. The intervention should ideally last two months.
  Assessments are conducted at 9 weeks of interval.

INTERVENTIONS:
Behavioral: Parental guidance — A psychological intervention including 4 sessions to assess how participants communicate with their children about the disease and take stock of their questions and difficulties. To identify children's reactions and needs. Practical situation are analyzed and worked through role play centered on communicational difficulties to enhance communicational self-efficacy and mutual support among participants. Emotional regulation strategies are learned through relaxation exercises. A relaxation booklet is given to the participants to practice at home too. Moreover, all participants receive an informational booklet containing age-appropriate recommendations on communication with children about cancer.
  Other Names: Efficacy of a parenting cancer related intervention
  Arms: Parental guidance

SUMMARY:
Background:

Cancer has a significant short and long-term impact on the family. Children of cancer patients may suffer from emotional, behavioral or somatic difficulties. Following the cancer diagnosis, many parents report being concerned about the impact of the illness on their children and how to communicate about the illness. In addition, they feel less able to meet the needs of their children and have difficulties regulating their emotions in response to their children's reactions.

Methods:

A randomized controlled trial was designed to assess the efficacy of a parental guidance intervention centered on communication with children in the context of a parental cancer.

This psychological intervention is designed to help parents and significant caregivers of the children. The participants are randomly assigned to either an intervention group (experimental group) or a waiting list group (control group).

The participants fill out self reported questionnaires that assess the parental self-efficacy in communication, mutual social support, communicational behaviors' with children, parenting concerns,communicational difficulties with children, knowledges about communication with children in oncological context, socio-demographical status, medical situation, psychiatric history, social difficulties and emotional state of the participants and children. The semi-structured interview with participants assesses their day to day communication with the children and the difficulties related to this communication. Those questionnaires are completed at baseline and post treatment (experimental group) and 9 weeks after baseline (control group).

This parental guidance consists of a weekly 4-session intervention. The aim of the sessions are to provide child support in the oncological context, mainly through communication.

Discussion:

This parental guidance would lead to improvements in knowledge, communication, parental self-efficacy and emotional regulation associated with child support.

DETAILED DESCRIPTION:
Introduction :

Parents raise many questions about the impact of the cancer on their children and on the communication with them about the disease. For many of them, the cancer impact their parental self-efficacy. This decrease of self-efficacy is related to difficulties to communicate openly with children and to regulate emotions in response to the feelings, reactions and questions of their children. In the same way, some parents report a lack of knowledge on how to support their children. They express doubts concerning the way they speak about cancer with their children.

Objectives of the study :

The primary objective of this study is to test the contribution and effectiveness of a psychological intervention in relation to the delivery of an informational booklet regarding participants' communication with the child in the oncology context. This intervention should increase participants' sense of communicative competence and communicationnal behaviors with children.

The secondary objectives is to evaluate the improvement of the participants' regarding the knowledge of how to support a child facing a parent's cancer, the emotional regulating capacity associated with participants' communication with the child, the evolution of the participants' concerns about the child. When the intervention is carried out in a dyad, it should also improve mutual support between participants.

This intervention is designed to help parents and significant caregivers of the children. It is focused on child support in the oncological context, and mainly on the communication between parents and their children. This intervention consists in a brief psychological intervention focused on improving knowledge, communication, parental self-efficacy and emotional regulation associated with child support. The intervention will be customized and tailored to each family.

Participants :

All significant caregivers of a child aged between 3 and 18 and who's facing parental cancer can be included in the study. A significant caregiver is a person who takes care of children at a practical, educational and emotional level (mostly parents, step parents, legal guardians, grandparents…). The whole study (assessment procedure and psychological intervention) is realized with one or two persons involved in child support. A consent form will be completed and signed by the adult participants.

Study design :

The effectiveness of the parental support intervention is assessed through a longitudinal two arms, randomized controlled trial. The psychological intervention is proposed to the main caregivers of children confronted to parental cancer.

In the experimental condition, the two significant caregivers of the child or the individual caregiver receive the intervention composed of an informational booklet and a psychological intervention. The intervention consists of four sessions, centered on supporting the child in the context of parental cancer mainly through communication.

In the control condition, the participants receive the informational booklet before being registered in a waiting list for the psychological intervention. The intervention should ideally last two months. Assessments are conducted at two periods (T1 and T2) : before and after the intervention for the experimental group and at 9 weeks of interval for the control group. The evaluation of the intervention is conducted through questionnaires completed by participants and a semi-structured interview.

Intervention :

The intervention consists in a brief psychological intervention including four sessions, centered on supporting the children in the context of parental cancer through communication. The content of the intervention is adapted to the specific situation of each family, their difficulties and their needs.

The first session is dedicated to the assessment of how participants communicate with their children about the disease and to take stock of their questions and difficulties. In this session, the family situation and the medical context are also discussed and the parental skills are identified. The other sessions are essentially focused on the identification of children's reactions and needs in the context of cancer and on the communication with children about the disease. Practical situation are analyzed and worked through role play centered on communicational difficulties. Participants must actively participate in the intervention. Specific techniques will be used with the participants to "co-construct" personalized communication with their child and to support its implementation. This active participation aims to enhance communicational self-efficacy and mutual support among participants. During the intervention, emotional regulation strategies are also transmitted to the participants through relaxation exercises in order to cope with the emotions felt in these particular contexts. A relaxation booklet is given to the participants to practice at home the relaxation exercises learned during the sessions. Moreover, all participants (experimental and control conditions) receive an informational booklet containing age-appropriate recommendations on communication with children about cancer. This booklet aims to improve knowledge of participants on how to support their children.

Assessment procedure :

Assessments are conducted at two periods (T1 and T2) and consist of questionnaires and a semi-structured interview with each participant. For the assessment, participants must refer specifically to only one child in their circle, aged between 3 and 18 years. If several children meet these criteria, participants determine the one for whom they have the most questions regarding communication with him/her about the illness. The child thus identified serves as a reference for T1 and T2 in order to standardize the evaluation procedure as much as possible.

Some questionnaires assess the primary outcome of the study : parental self-efficacy in communication, communicational behaviors' with children. Other questionnaires assess the secondary outcome of the study: Emotional regulation, mutual support between participants, communicationnal difficulties with children, parenting concerns, knowledges about communication with children in oncological context. Many questionnaires are specifically created by the investigator's team. Other questionnaires assess control variables: the socio-demographical status, medical situation, psychiatric history, social difficulties and emotional state of the participants and children. The semi-structured interview with participants assesses their day to day communication with the children and the difficulties related to this communication. Each semi-structured interview takes approximatively 20 minutes and is recorded and transcribed.

The sample size has been calculated a priori in order to detect the differences in the evolution of the two groups (experimental and control conditions) between T1 and T2.

The sample size calculation was done with the software G*Power. The power analysis has been based on a previous pilot study assessing the efficacy of the intervention on patient. Self-efficacy score have been considered to perform the power analysis (Change over time in Experimental Group: Delta T2-T1 Mean = 0.9514; SD = 0.8043; Change over time Control Group is consider as zero). The effect size was 1.183 for a power of 0.90 in two-side. Based on this result but considering the small sample of the pilot study, the sample size calculation has been based on a 0.9% power, an effect-size of 0.9 and a two-sided α = 0.05 t-test. Considering this power analysis, 54 evaluable patients are therefore needed for the efficacy assessment. Considering a drop-out rate of approximately 10%, 6 patients should be moreover recruited. The aim of the study is therefore to recruit 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Significant caregiver of a child aged between 3 and 18 who's facing parental cancer
* Participants must be of legal age
* Participants must not have an acute psychiatric or neurological disorder
* Participants must have sufficient command of French (speaking, writing, reading)
* Completing a written informed consent

Exclusion Criteria:

* Pre-terminal or terminal stage of cancer of the parent
* Death of the parent

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Change of the parental self-efficacy in communication | 8-9 weeks
  Assessment through a self-reported scale created for the study and completed by the participants named "Sense of communicational competence with the child". The questionnaire is composed of 16 items. The scale represents the level of certainty regarding the proposed items. The questionnaire has a 10 points Likert scale. The scale ranges is from 0 to 10. 0 means " not at all certain " and 10 "quite certain". Change in the parental self-efficacy in communication is assessed by comparing the questionnaire completed in T1 with the one completed in T2.
  Parental self-efficacy is also analyzed through a content analysis of the responses given by the participants in the semi-structured interview. The presence of words such as confident, capable or opposite will provide insight into the sense of parental self-efficacy. Comparing the responses in T1 with those in T2 will highlight the change of parental self-efficacy through the increase or decrease in the occurrence of a word.
Change of the communicational behavior | 8-9 weeks
  Assessment through a content analysis of the responses given by the participants in the semi-directive interview. The main domains explore by the semi directive interview are: description of the communication, feelings during the communication and communicational behaviors. Comparing the responses in T1 with those in T2 will highlight the evolution of the communicational behaviors with the child.

SECONDARY OUTCOMES:
Evaluation of the Emotional distress | 8-9 weeks
  Assessed through a validated self-reported scale: The Hospital Anxiety and Depression Scale (HADS). It is composed by two dimensions (anxiety and depression) and has a 4 point Likert scale that vary at each item. HADS provides a total score (0-42 range) by summing all item scores. A higher score reflects a higher emotional distress. Anxiety subscale score (0-21 range) is provided by summing all Anxiety-items. A higher score reflects more anxiety. Depression subscale scores (0-21 range) is provided by summing all Depression-items. A higher score reflects more depression.
Evaluation of the Communicationnal difficulties with the child | 8-9 weeks
  Communicational difficulties are assessed through a self-reported scale created for the study and completed by the participants named "Communication difficulties with the child ". The scale is composed of 13 items which represents the level of truth regarding the proposed items. The questionnaire has a 4 points Likert scale. The scale ranges is from "yes" to "no ". The evolution of the communicational difficulties is assessed by comparing the questionnaire completed in T1 with the one completed in T2.
Description of the Communicationnal difficulties with the child | 8-9 weeks
  The Communicational difficulties with children are also analysed through a content analysis of the responses given by the participants in the semi-directive interview. The main domains explore by the semi directive interview are: description of the communication, feelings during the communication and communicational behaviors. Comparing the responses in T1 with those in T2 will highlight the evolution of the communicational difficulties.
Evaluation of the mutual support between participants | 8-9 weeks
  Mutual support between participants is assessed through a self-reported scale created for the study and completed by the participants named "Mutual support between participants". The scale is composed of 8 items which represents the level of truth regarding the proposed items. The questionnaire has a 4 points Likert scale. The scale ranges is from "yes" to "no". The evolution of the mutual support between participants is assessed by comparing the questionnaire completed in T1 with the one completed in T2.
Evaluation of parenting concerns | 8-9 weeks
  Parents' concerns are assessed through a self-reported scale created for the study and completed by the participants named "concerns about the identified child". The scale is composed of 14 items which represents the level of truth regarding the proposed items. The questionnaire has a 5 points Likert scale. The scale ranges is from "Not at all concerned" to "deeply concerned". The evolution of parenting concerns is assessed by comparing the questionnaire completed in T1 with the one completed in T2.
Evaluation of the knowledges of the participant about the understanding of children in oncological context | 8-9 weeks
  Assessment through a self-reported scale created for the study and completed by the participants named "Knowledge of the child's level of understanding about cancer". It is composed by 10 items that describe a child's ability to understand cancer disease. The questionnaire has a 2 points Likert scale, "yes" or "no". The expected answers are 6 yes and 4 no. The answers will show the level of knowledge of the participant (good, medium or bad) regarding the understanding of children. The evolution of the knowledges of the participant about the understanding of children in oncological context is assessed by comparing the questionnaire completed in T1 with the one completed in T2.

CONTACTS AND LOCATIONS:
Overall Officials: Razavi, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauch PK, Muriel AC. The importance of parenting concerns among patients with cancer. Crit Rev Oncol Hematol. 2004 Jan;49(1):37-42. doi: 10.1016/s1040-8428(03)00095-7. PMID 14734153
- [Result] Cessna JM, Pidala J, Jacobsen PB. Relationships between parenting self-efficacy and distress in parents who have school-aged children and have been treated with hematopoietic stem cell transplant or have no cancer history. Psychooncology. 2016 Mar;25(3):339-46. doi: 10.1002/pon.3848. Epub 2015 May 12. PMID 25967755
- [Result] Ellis SJ, Wakefield CE, Antill G, Burns M, Patterson P. Supporting children facing a parent's cancer diagnosis: a systematic review of children's psychosocial needs and existing interventions. Eur J Cancer Care (Engl). 2017 Jan;26(1). doi: 10.1111/ecc.12432. Epub 2016 Jan 18. PMID 26776913
- [Result] Huizinga GA, Visser A, Zelders-Steyn YE, Teule JA, Reijneveld SA, Roodbol PF. Psychological impact of having a parent with cancer. Eur J Cancer. 2011 Sep;47 Suppl 3:S239-46. doi: 10.1016/S0959-8049(11)70170-8. No abstract available. PMID 21943981
- [Result] Inhestern L, Haller AC, Wlodarczyk O, Bergelt C. Psychosocial Interventions for Families with Parental Cancer and Barriers and Facilitators to Implementation and Use - A Systematic Review. PLoS One. 2016 Jun 8;11(6):e0156967. doi: 10.1371/journal.pone.0156967. eCollection 2016. PMID 27276079
- [Result] Koopman HM, Baars RM, Chaplin J, Zwinderman KH. Illness through the eyes of the child: the development of children's understanding of the causes of illness. Patient Educ Couns. 2004 Dec;55(3):363-70. doi: 10.1016/j.pec.2004.02.020. PMID 15582342
- [Result] Kuhl PK. Early language acquisition: cracking the speech code. Nat Rev Neurosci. 2004 Nov;5(11):831-43. doi: 10.1038/nrn1533. PMID 15496861
- [Result] Lewis FM, Brandt PA, Cochrane BB, Griffith KA, Grant M, Haase JE, Houldin AD, Post-White J, Zahlis EH, Shands ME. The Enhancing Connections Program: a six-state randomized clinical trial of a cancer parenting program. J Consult Clin Psychol. 2015 Feb;83(1):12-23. doi: 10.1037/a0038219. Epub 2014 Nov 17. PMID 25403016
- [Result] Merckaert I, Libert Y, Lieutenant F, Moucheux A, Farvacques C, Slachmuylder JL, Razavi D. Desire for formal psychological support among caregivers of patients with cancer: prevalence and implications for screening their needs. Psychooncology. 2013 Jun;22(6):1389-95. doi: 10.1002/pon.3153. Epub 2012 Aug 8. PMID 22888079
- [Result] Merckaert I, Libert Y, Messin S, Milani M, Slachmuylder JL, Razavi D. Cancer patients' desire for psychological support: prevalence and implications for screening patients' psychological needs. Psychooncology. 2010 Feb;19(2):141-9. doi: 10.1002/pon.1568. PMID 19382112
- [Result] Moore CW, Rauch PK, Baer L, Pirl WF, Muriel AC. Parenting changes in adults with cancer. Cancer. 2015 Oct 1;121(19):3551-7. doi: 10.1002/cncr.29525. Epub 2015 Jun 19. PMID 26094587
- [Result] Muriel AC, Moore CW, Baer L, Park ER, Kornblith AB, Pirl W, Prigerson H, Ing J, Rauch PK. Measuring psychosocial distress and parenting concerns among adults with cancer: the Parenting Concerns Questionnaire. Cancer. 2012 Nov 15;118(22):5671-8. doi: 10.1002/cncr.27572. Epub 2012 Apr 19. PMID 22517236
- [Result] Niemela M, Paananen R, Hakko H, Merikukka M, Gissler M, Rasanen S. The prevalence of children affected by parental cancer and their use of specialized psychiatric services: the 1987 Finnish Birth Cohort study. Int J Cancer. 2012 Nov 1;131(9):2117-25. doi: 10.1002/ijc.27466. Epub 2012 Mar 22. PMID 22307957
- [Result] Paradis M, Consoli SM, Pelicier N, Lucas V, Andrieu JM, Jian R. [Psychosocial distress and communication about cancer in ill partners and their spouses]. Encephale. 2009 Apr;35(2):146-51. doi: 10.1016/j.encep.2008.02.008. Epub 2008 Jun 13. French. PMID 19393383
- [Result] Semple CJ, McCaughan E. Family life when a parent is diagnosed with cancer: impact of a psychosocial intervention for young children. Eur J Cancer Care (Engl). 2013 Mar;22(2):219-31. doi: 10.1111/ecc.12018. Epub 2012 Dec 12. PMID 23231498
- [Result] Syse A, Aas GB, Loge JH. Children and young adults with parents with cancer: a population-based study. Clin Epidemiol. 2012;4:41-52. doi: 10.2147/CLEP.S28984. Epub 2012 Mar 13. PMID 22442635

DOCUMENTS (1):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03905278/Prot_000.pdf